CLINICAL TRIAL: NCT00804674
Title: Improved Pain Relief Using Intermittent Bupivacain Injections at the Donor Site After Breast Reconstruction With Deep Inferior Epigastric Artery Perforator (DIEP) Flap
Brief Title: Pain Study Using Intermittent Bupivacain Injections After Breast Reconstruction With DIEP Flap
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Responsible Party: Jørgen Utvoll MD, ullevaal university hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 01
Record Dates: First submitted 2008-12-03; First posted 2008-12-09 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-06

CONDITIONS: Breast Reconstruction
Keywords: bupivacain; breast; reconstruction; diep; pain; postoperative; catheter; anesthesia
MeSH Terms: conditions — Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 bupivacain (Active Comparator)
  Interventions: Drug: bupivacain
- 2 placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: bupivacain
  Arms: 1 bupivacain
Drug: placebo
  Arms: 2 placebo

SUMMARY:
patients are given bupivacain intermittent locally on the donor site after brest reconstruction with diep flap. The hypothesis was that this approach will reduce the need for rescue analgetic medication and pain perception within the three first days

ELIGIBILITY:
Inclusion Criteria:

* all patients planned to undergo reconstructive breast surgery with a DIEP

Exclusion Criteria:

* regular use of analgesics
* known allergic reaction to bupivacain
* bleeding disorders
* pregnancy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-08; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: jørgen utvoll, MD, Principal Investigator — Consultant at ullevaal university hospital